CLINICAL TRIAL: NCT05891197
Title: A Biomarker Screening Protocol to Support Preliminary Eligibility for Clinical Trials Evaluating Safety and Efficacy of Adoptive T-cell Therapies in Participants With Solid Tumors
Brief Title: A Biomarker Screening Protocol for Participants With Solid Tumors
Acronym: START
Status: Terminated | Type: Observational
Why Stopped: Pipeline Reprioritization
Sponsor: Lyell Immunopharma, Inc. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: LYLSCR-101
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Triple Negative Breast Cancer; Non-small Cell Lung Cancer; Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Metastatic; Non-Small Cell Carcinoma of Lung, TNM Stage 4; Advanced Breast Cancer; Advanced Lung Carcinoma; NSCLC; NSCLC, Recurrent; NSCLC Stage IV; Relapsed Cancer; Relapse/Recurrence; Recurrent Breast Cancer; Recurrent NSCLC; Platinum-resistant Ovarian Cancer; Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer; Endometrial Cancer; Endometrioid Tumor; High Grade Serous Carcinoma; Ovarian Epithelial Cancer
Keywords: Biomarker Screening; Immunotherapy; CAR-T; CAR T-cell therapy; CAR T; CAR T-cell; ROR1; ROR1+; ROR1 positive; cell therapy; relapsed; refractory; solid tumor; advanced; metastatic; breast cancer; lung cancer; triple negative breast cancer; non small cell lung cancer; ovarian cancer; endometrial cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Recurrence; Breast Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Carcinoma, Ovarian Epithelial; Neoplasm Metastasis; Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — An Archival tumor tissue sample collected within 3 years prior to enrollment. The sample must consist, at minimum, of 5 freshly cut, unstained 4-5 μM sections cut from a formalin-fixed paraffin-embedded (FFPE) tissue block. The sample must contain sufficient tumor tissue to allow for the evaluation of biomarker expression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Biomarker Screening Protocol for Preliminary Eligibility Determination for Adoptive T-cell Therapy Trials:This is a decentralized, multi-site, US-based biomarker screening study to identify participants who have specific disease indications and tumor expression of target(s) of interest that may inform eligibility for active and future Lyell clinical trials. No investigational treatments will be administered in this non-interventional screening study. Only previously obtained archival tumor tissue will be allowed on this study for biomarker analysis. Fresh tumor biopsies are not permitted on this study. The study will be conducted virtually and participants will utilize telehealth and e-consent modules. If participants tumors express the biomarkers of interest they can be referred to open and enrolling clinical trials. Participation on the screening study does not guarantee enrollment or treatment on an interventional clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged ≥ 18 years at time of informed consent
2. Able to provide informed consent
3. Histologically or cytologically confirmed diagnosis of advanced or metastatic solid tumor malignancy.The Sponsor will indicate which solid tumor disease indications are open to enrollment.
4. Ability to provide a tumor tissue sample collected within 3 years prior to enrollment. The sample must consist, at minimum, of 5 freshly cut, unstained 4-5 μM sections cut from a formalin-fixed paraffin-embedded (FFPE) tissue block. The sample must contain sufficient tumor tissue to allow for the evaluation of biomarker expression

Exclusion Criteria:

1. Prior solid organ transplantation
2. Prior treatment with any adoptive cell therapy
3. Uncontrolled medical, psychological, familial, sociological, or geographical conditions that do not permit compliance with a clinical study, as judged by the Investigator or Sponsor's Medical Monitor

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 years of age or older with histologically or cytologically confirmed diagnosis of advanced or metastatic solid tumor malignancy who are willing to have archival tumor tissue analyzed for biomarker(s).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
To identify participants whose tumors express biomarkers, such as ROR1, that may inform eligibility for active and future Lyell clinical trials | 5 years

SECONDARY OUTCOMES:
To explore tumor expression of biomarkers, such as ROR1, by different methods (e.g., IHC versus next-generation sequencing [NGS]) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Walling, MBChB, PhD, Study Chair — Lyell Immunopharma
Locations (1):
- Accellacare, Rocky Mount, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided